CLINICAL TRIAL: NCT00997373
Title: Predicting Aromatase Inhibitor Responsiveness in Endometrial Carcinoma
Brief Title: Letrozole as a Treatment of Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200917341; CFEM 345AUS63
Record Dates: First submitted 2009-10-15; First posted 2009-10-19 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Endometrial Carcinoma
Keywords: Endometrial Cancer; Endometrial Carcinoma; Aromatase Inhibitor; Letrozole; Femara
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Letrozole (Experimental): letrozole 2.5 mg PO daily for 2-3 weeks prior to hysterectomy.
  Interventions: Drug: Letrozole
- control (No Intervention): no treatemtn prior to hysterectomy

INTERVENTIONS:
Drug: Letrozole — 2.5 mg daily from the day of enrollment to the day before surgery, generally about 3 weeks
  Other Names: Femara; 4-[(4-cyanophenyl)-(1,2,4-triazol-1-yl)methyl]benzonitrile,; CAS number 112809-51-5
  Arms: Letrozole

SUMMARY:
Some cases of endometrial cancer are dependent on estrogen for their growth. Letrozole blocks estrogen production in the body. The purpose of this study is to determine if the investigators can predict which patients might benefit from Letrozole treatment by studying the many different forms of the estrogen receptor molecule that exist within the cancer tissues. To participate in this study, the patients must be 40 years of age or older and have biopsy-proven endometrial carcinoma, either well differentiated or moderately differentiated forms. Also, to be eligible to participate in this study, the patients need to be healthy enough to have a hysterectomy. If the patients are less than age 60, they will need a blood test (FSH) to confirm that they have gone into menopause.

ELIGIBILITY:
Inclusion Criteria:

* FIGO grade 1 or 2 endometrioid adenocarcinoma of the endometrium
* Post menopausal status must be demonstrated
* Signed informed consent

Exclusion Criteria:

* FIGO grade 3 endometrioid adenocarcinoma or non-endometrioid cancers of the endometrium
* Younger than 40 or postmenopausal status not established
* Pregnant or breastfeeding

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lloyd H. Smith, MD, PhD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California Davis, Sacramento, California
  - University of California, Davis, Sacramento, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment by providing gynecologic oncologist beginning 11/2/2009
Pre-assignment Details: Non-randomized selection of control subjects
Groups:
- Letrozole: Letrozole 2.5 mg PO daily for 2-3 weeks prior to hysterectomy or re-biopsy.
  Letrozole: 2.5 mg daily from the day of enrollment to the day before surgery (generally about 3 weeks) or to the day of repeat endometrial biopsy 9medical treatment arm).
- Control: No treatment prior to hysterectomy
Period: Overall Study
Arm/Group | Letrozole | Control
Started | 28 | 15
Received Letrozole | 23 | 0
Completed Hysterectomy | 17 | 15
Completed | 13 | 15
Not Completed | 15 | 0
Not completed — Withdrawal by Subject | 5 | 0
Not completed — wrong tumor type | 4 | 0
Not completed — could not have hysterectomy | 6 | 0

BASELINE CHARACTERISTICS:
Population: Subjects and controls selected to give groups similar in age and tumor grade. Four subjects excluded - wrong tumor type. One treatment arm completed but was excluded from analysis because of late completion.
Groups:
- Letrozole Arm: Grade 1 or 2 endometrial cancer treated 3 weeks before hysterectomy of repeat biopsy. Letrozole 2.5 mg PO daily.
- Control: No letrozole before hysterectomy
- Total: Total of all reporting groups
Arm/Group | Letrozole Arm | Control | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Changes in Ki67 Expression After About 3 Weeks of Letrozole Treatment for Patients With Endometrial Cancer
Description: Changes in %Ki67 staining cells by immunoperoxidase of paraffin embedded, formalin fixed tissue
Time Frame: At time of consent and after hysterectomy (generally about 3 weeks)
Population: Subjects completing treatment who had confirmed histopathology compared to a non-randomized group of untreated control subjects. "Aromatase inhibitor responsiveness" was defined as a proportionate decline in %Ki67 staining of at least 70% between pre-treatment biopsy and hysterectomy 9or repeat biopsy).
Measure: Mean (Full Range); unit: percentage of Ki67 staining cells
Arm/Group | Letrozole | Control
Number analyzed (Participants) | 12 | 12
percentage of Ki67 staining cells | -3.75 [-18 to 24] | 1.583 [-30 to 21]
Statistical Analysis 1: Comparison: Letrozole vs Control; Test type: Superiority or Other; p = 0.0373, Fisher Exact

ADVERSE EVENTS:
Time Frame: Weekly by telephone interview during treatment
Description: Adverse events for control arm not collected.
Arm/Group | Letrozole | Control
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/0
Other Adverse Events (participants affected / at risk) | 3/23 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole (N=23) | Control (N=0)
death (Cardiac disorders) | 1 (1) | 0 (0) — Subject with severe pre-existing pulmonary hypertension expired at home suddenly of apparent acute cardiac event 2 weeks after starting letrozole.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole (N=23) | Control (N=0)
fatigue (General disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No